CLINICAL TRIAL: NCT02700451
Title: A Randomized Controlled Trial of Post-operative Acetaminophen Versus Nonsteroidal Anti-Inflammatory Drug (NSAID) Use on Lumbar Spinal Fusion Outcomes
Brief Title: Post-op Acetaminophen vs NSAID Use on Lumbar Spinal Fusion Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-333
Record Dates: First submitted 2016-02-18; First posted 2016-03-07 (Estimated); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Lumbar Osteoarthritis; Spondylosis; Lumbar Disc Disease; Spinal Stenosis
Keywords: IV acetaminophen; IV Ketorolac; Post-operative analgesia; Opioid use
MeSH Terms: conditions — Osteoarthritis, Spine; Spondylosis; Intervertebral disc disease; Spinal Stenosis | interventions — Ketorolac; Ketorolac Tromethamine; Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravenous (IV) Placebo (Placebo Comparator): IV Placebo arm
  Interventions: Drug: Placebo
- IV Ketorolac (Experimental): IV Ketorolac arm
  Interventions: Drug: Ketorolac
- IV Acetaminophen (Experimental): IV Acetaminophen arm
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Ketorolac — Age 18-64: Intravenous Ketorolac 30 milligrams (mg) every 6 hours for 48 hours in addition to patient-controlled analgesia and oral opioids as needed.
  Age 65-75: Intravenous Ketorolac 15 milligrams (mg) every 6 hours for 48 hours in addition to patient-controlled analgesia and oral opioids as needed.
  Other Names: Toradol
  Arms: IV Ketorolac
Drug: Acetaminophen — Intravenous Acetaminophen 1000mg every 6 hours for 48 hours in addition to patient-controlled analgesia and oral opioids as needed.
  Other Names: Tylenol, Ofirmev
  Arms: IV Acetaminophen
Drug: Placebo — Intravenous Normal Saline every 6 hours for 48 hours in addition to patient-controlled analgesia and oral opioids as needed.
  Other Names: Normal Saline
  Arms: Intravenous (IV) Placebo

SUMMARY:
Patients undergoing spine surgery often have considerable pain post-operatively and frequently require opioid medication (Percocet, Norco, oxycodone, morphine, etc.) to control their pain postoperatively. The widespread use of opioids, however, is associated with a number of side effects. These include: sedation, dizziness, nausea, vomiting, constipation, dizziness and itching amongst others. Some investigators have suggested that anti-inflammatory medications (the same class of medicines as advil, ibuprofen, etc.) and acetaminophen (Tylenol) can reduce the total dose of opioid required postoperatively and, as a result, lower opioid-related side effects.

The purpose of this study is to test this hypothesis and determine if postoperative anti-inflammatory medications and postoperative acetaminophen can reduce the amount of opioid required to control pain following surgery. A secondary goal of this study is to examine if the change in pain medication will lead to decreased overall pain levels, decreased opioid-related side effects and improved function [quicker ambulation with physical therapy (PT), earlier return to work, etc.].

DETAILED DESCRIPTION:
Given the potential for non-steroidal anti inflammatory drugs (NSAIDs) and acetaminophen to decrease opioid requirements following spine surgery, the investigators propose a prospective, randomized, double-blinded clinical trial comparing the efficacy of intravenous (IV) acetaminophen (Group A) or IV ketorolac (Group K) versus placebo (Group P). The impact of treatment on perioperative opioid use, opioid-related complications, functional outcomes and rates of pseudarthrosis following 1 or 2 level lumbar fusion surgery will be measured in each group. The specific aims of this study are as follows:

* Specific Aim 1: Determine the impact of IV ketorolac or IV acetaminophen use on immediate postoperative opioid requirements, postoperative pain levels and opiate related symptoms using the Opiate-Related Symptom Distress Scale (ORSDS)
* Specific Aim 2: Determine the impact of IV ketorolac or IV acetaminophen use on functional outcomes defined by return to work, Oswestry Disability Index (ODI) and the Veterans Rand-12 (VR-12) Health Survey

The primary outcome is to determine the total postoperative opioid dose (in oral morphine equivalents) in each group. The investigators hypothesize that patients in Group A and Group K will have lower total opioid use, suffer from fewer opiate related symptoms and have similar rates of pseudarthrosis to patients in Group P. The investigators hypothesize that patients in Group A and Group K will have a quicker return to work and improved early functional outcomes although they acknowledge that long term functional outcomes may be the same for all groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Require 1 or 2 level lumbar spinal fusion through posterior or lateral approach
* No history of long term opioid use (daily or almost daily opioid use > 2 weeks) and not on opiates at time of presentation to clinic

Exclusion Criteria:

* Documented allergy to NSAIDs or Acetaminophen
* History of: Peptic Ulcer Disease, Congestive heart failure, Chronic liver disease, Elevated alanine aminotransferase (ALT)/ aspartate aminotransferase (AST) greater than 1.5 times control, Bleeding disorder, Renal dysfunction (Serum creatinine > 1.5 mg/dL), Glucocorticoid use within 1 month of surgery
* Current smokers (quite date < 30 days ago)
* Revision for pseudarthrosis
* Patients who are unable to physically or mentally provide consent to the study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2016-03; Primary Completion 2021-12-31 (Actual); Study Completion 2023-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Himo Gang, Study Director — Research Manager for Spine Research; Harvinder Sandhu, MD, Principal Investigator — Associate Professor of Orthopedic Surgery
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Assessed for eligibility (n= 1,372) Excluded (n= 1,194)
  * Not meeting inclusion criteria (n= 1,137)
  * Declined to participate (n= 132)
  * Other reasons (n= 103)
Groups:
- IV Ketorolac: IV Ketorolac arm
  Ketorolac: Age 18-64: Intravenous Ketorolac 30 milligrams (mg) every 6 hours for 48 hours in addition to patient-controlled analgesia and oral opioids as needed.
  Age 65-75: Intravenous Ketorolac 15 milligrams (mg) every 6 hours for 48 hours in addition to patient-controlled analgesia and oral opioids as needed.
Period: Overall Study
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Started | 60 | 60 | 58
Completed | 44 | 43 | 41
Not Completed | 16 | 17 | 17
Not completed — Protocol Violation | 2 | 2 | 3
Not completed — Discontinued intervention | 14 | 15 | 14

BASELINE CHARACTERISTICS:
Population: Analysis performed on Per-Protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen | Total
Number analyzed (Participants) | 44 | 43 | 41 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 32 | 31 | 94
  >=65 years | 13 | 11 | 10 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (11.2) | 56.3 (11.1) | 56.1 (13.2) | 57.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 20 | 55
  Male | 26 | 26 | 21 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 44 | 40 | 39 | 123
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 44 | 43 | 41 | 128

OUTCOME MEASURES:

1. Primary Outcome: Perioperative Opioid Use
Description: Measure the impact of treatment on total opioid use during the hospital stay
Time Frame: Hospital stay (2-4 days)
Measure: Median (Inter-Quartile Range); unit: oral morphine equivalents (OME) (mmg)
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 44 | 43 | 41
oral morphine equivalents (OME) (mmg)
  OME total in the first 72H | 86.25 [39.6 to 245.55] | 306.6 [161 to 423] | 192.4 [91.55 to 372.85]
  OME total to discharge | 88.95 [46.2 to 284.03] | 324 [169 to 471] | 237.9 [91.55 to 467.05]
Statistical Analysis 1: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of OME total in the first 72H is the same across these arms; Test type: Equivalence — Two-sided 95% confidence interval; p < 0.001, Kruskal-Wallis — Threshold for statistical significance was p = 0.05
Statistical Analysis 2: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of OME total to discharge is the same across these arms; Test type: Equivalence — Two-sided 95% confidence interval; p < 0.001, Kruskal-Wallis — The thresholds for statistical significant was p = 0.05

2. Secondary Outcome: Opioid Use at 4-6 Weeks
Description: Track opioid use after discharge for the first 4-6 weeks
Time Frame: 4-6 weeks
Population: Patient treated Per-Protocol with completed follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 43 | 39 | 36
Participants
  No opioid use | 34 | 33 | 22
  Opioid use | 9 | 6 | 14
Statistical Analysis 1: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; Similar Distribution of opioid use between the 3 arms; Test type: Equivalence — Two-sided; p = 0.048, Chi-squared

3. Secondary Outcome: Opioid Use at 3 Months
Description: Track opioid use after discharge for the first 3 months; assess for continued opioid use
Time Frame: 3 months
Population: Patient treated Per-Protocol with completed follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 37 | 27 | 31
Participants
  No opioid use | 32 | 25 | 26
  Opioid use | 5 | 2 | 5
Statistical Analysis 1: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; Test type: Equivalence — Two-sided; p = 0.595, Chi-squared

4. Secondary Outcome: Opioid Use at 1 Year
Description: Track opioid use after discharge for the first 1 year; assess for continued opioid use
Time Frame: 1 year
Population: Patient treated Per-Protocol with completed follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 33 | 31 | 22
Participants
  No opioid use | 32 | 31 | 21
  Opioid use | 1 | 0 | 1

5. Secondary Outcome: Opioid Use at 2 Years
Description: Track total opioid use after discharge for the first 2 years; assess for continued opioid use
Time Frame: 2 years
Population: Patient treated Per-Protocol with completed follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 27 | 27 | 25
Participants
  No opioid use | 26 | 26 | 22
  Opioid use | 1 | 1 | 3

6. Secondary Outcome: Numerical Pain Rating Scale
Description: Validated pain scale; will be completed by patient Minimum Score: 0 & Maximum score 100 A lower score is representative of a low pain level
Time Frame: 1 days and 3 days
Population: Analysis performed on patient with data completed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 44 | 43 | 41
units on a scale
  POD1 - Current pain level: number analyzed (Participants) | 27 | 28 | 29
  POD1 - Current pain level | 39 [22 to 58] | 46 [29.3 to 72] | 42 [25.5 to 67]
  POD1 - Best pain level: number analyzed (Participants) | 27 | 28 | 29
  POD1 - Best pain level | 23 [13 to 40] | 24.5 [13 to 34.5] | 21 [12.5 to 51]
  POD1 - Worst pain level: number analyzed (Participants) | 27 | 28 | 29
  POD1 - Worst pain level | 62 [44 to 73] | 89.5 [66.3 to 97.8] | 74 [54 to 86.5]
  POD3 - Current pain level: number analyzed (Participants) | 20 | 21 | 20
  POD3 - Current pain level | 66 [26 to 76.8] | 47 [25.5 to 74] | 52 [25 to 65.0]
  PDO3 - Best pain level: number analyzed (Participants) | 19 | 21 | 20
  PDO3 - Best pain level | 23 [12 to 36] | 25 [12.5 to 50] | 39 [18.8 to 51]
  POD3 - Worst pain level: number analyzed (Participants) | 19 | 21 | 41
  POD3 - Worst pain level | 84 [69 to 88] | 83 [51.5 to 93.5] | 72.5 [62.8 to 85]
Statistical Analysis 1: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD1 - Current pain level is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.732, Kruskal-Wallis
Statistical Analysis 2: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD1 - Best pain level is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.896, Kruskal-Wallis
Statistical Analysis 3: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD1 - Worst pain level is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.004, Kruskal-Wallis
Statistical Analysis 4: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD3 - Current pain level is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.325, Kruskal-Wallis
Statistical Analysis 5: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD3 - Best pain level is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.283, Kruskal-Wallis
Statistical Analysis 6: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD3 - Worst pain level is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.610, Kruskal-Wallis

7. Secondary Outcome: Brief Pain Inventory
Description: The Brief Pain Inventory (BPI) is a self-administered questionnaire for chronic pain conditions. The BPI gives two main scores: a pain severity score and a pain interference score. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40. The pain interference score corresponds to the item on pain interference. The seven sub-items are rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score, ranging from 0 to 70. The first item, pain drawing diagrams (painful and most painful areas) and the items on pain relief treatment or medication (list of the treatments and amount of relief) do not contribute to the scoring.
Time Frame: 1 day and 3 days
Population: Patient treated Per-Protocol with completed follow-up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 44 | 43 | 41
score on a scale
  POD1 - Pain has interfered with General Activity: number analyzed (Participants) | 44 | 40 | 38
  POD1 - Pain has interfered with General Activity | 6.5 [3.25 to 10] | 9 [6 to 10] | 9 [6 to 10]
  POD1 - Pain has interfered with Mood: number analyzed (Participants) | 44 | 39 | 38
  POD1 - Pain has interfered with Mood | 2 [0 to 6] | 4 [0 to 6] | 1.5 [0 to 6]
  POD1 - Pain has interfered with Walking Ability: number analyzed (Participants) | 43 | 40 | 38
  POD1 - Pain has interfered with Walking Ability | 5 [2 to 9] | 7 [5.25 to 10] | 7 [5 to 9]
  POD1 - Pain has interfered with Normal work: number analyzed (Participants) | 42 | 38 | 37
  POD1 - Pain has interfered with Normal work | 8 [3.75 to 10] | 10 [7 to 10] | 8 [6.5 to 10]
  POD1 - Pain has interfered with Relation with other: number analyzed (Participants) | 44 | 40 | 38
  POD1 - Pain has interfered with Relation with other | 0 [0 to 3.75] | 2.5 [0 to 5.75] | 1.5 [0 to 6]
  POD1 - Pain has interfered with Sleep: number analyzed (Participants) | 44 | 40 | 38
  POD1 - Pain has interfered with Sleep | 3 [1 to 6.75] | 5 [1 to 8.75] | 6 [2.75 to 8]
  POD1 - Pain has interfered with Enjoyment of life: number analyzed (Participants) | 44 | 40 | 38
  POD1 - Pain has interfered with Enjoyment of life | 5 [2 to 8.75] | 9 [5 to 10] | 7 [4 to 10]
  POD3 - Pain has interfered with General Activity: number analyzed (Participants) | 35 | 35 | 29
  POD3 - Pain has interfered with General Activity | 8 [3 to 10] | 7 [5 to 10] | 8 [7 to 10]
  POD3 - Pain has interfered with Mood: number analyzed (Participants) | 35 | 36 | 29
  POD3 - Pain has interfered with Mood | 5 [1 to 7] | 3 [0 to 6.75] | 5 [2 to 7]
  POD3 - Pain has interfered with Walking Ability: number analyzed (Participants) | 35 | 36 | 29
  POD3 - Pain has interfered with Walking Ability | 5 [4 to 7] | 4.5 [3 to 8] | 6 [5 to 7]
  POD3 - Pain has interfered with Normal work: number analyzed (Participants) | 35 | 36 | 28
  POD3 - Pain has interfered with Normal work | 9 [8 to 10] | 10 [5.25 to 10] | 8 [6.25 to 10]
  POD3 - Pain has interfered with Relation with other: number analyzed (Participants) | 35 | 36 | 29
  POD3 - Pain has interfered with Relation with other | 2 [0 to 7] | 2 [0 to 5] | 4 [0 to 6]
  POD3 - Pain has interfered with Sleep: number analyzed (Participants) | 35 | 36 | 28
  POD3 - Pain has interfered with Sleep | 6 [4 to 8] | 4 [1.25 to 7] | 5 [4 to 7.75]
  POD3 - Pain has interfered with Enjoyment of life: number analyzed (Participants) | 35 | 36 | 29
  POD3 - Pain has interfered with Enjoyment of life | 7 [4 to 9] | 6.5 [3.25 to 10] | 8 [5.5 to 9]
Statistical Analysis 1: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD1 - Pain has interfered with General Activity is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.016, Kruskal-Wallis
Statistical Analysis 2: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD1 - Pain has interfered with Mood is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.294, Kruskal-Wallis
Statistical Analysis 3: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD1 - Pain has interfered with Walking Ability is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.016, Kruskal-Wallis
Statistical Analysis 4: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD1 - Pain has interfered with Normal work is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.082, Kruskal-Wallis
Statistical Analysis 5: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD1 - Pain has interfered with Relation with other is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.117, Kruskal-Wallis
Statistical Analysis 6: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD1 - Pain has interfered with Sleep is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.061, Fisher Exact
Statistical Analysis 7: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD1 - Pain has interfered with Enjoyment of life is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.023, Kruskal-Wallis
Statistical Analysis 8: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD3 - Pain has interfered with General Activity is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.681, Kruskal-Wallis
Statistical Analysis 9: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD3 - Pain has interfered with Mood is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.405, Kruskal-Wallis
Statistical Analysis 10: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD3 - Pain has interfered with Walking Ability is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.458, Kruskal-Wallis
Statistical Analysis 11: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD3 - Pain has interfered with Normal work is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.482, Kruskal-Wallis
Statistical Analysis 12: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD3 - Pain has interfered with Relation with other is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.544, Kruskal-Wallis
Statistical Analysis 13: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD3 - Pain has interfered with Sleep is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.202, Kruskal-Wallis
Statistical Analysis 14: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of POD3 - Pain has interfered with Enjoyment of life is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.580, Kruskal-Wallis

8. Secondary Outcome: Opioid Related Side Effects
Description: Ileus, nausea/vomiting, first bowel movement, first flatus, treated pruritis will be identified and recorded
Time Frame: Hospital Stay (1-4 days)
Population: Patient treated Per-Protocol with completed follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 44 | 43 | 41
Participants
  POD1 - Nausea?: number analyzed (Participants) | 44 | 40 | 38
  POD1 - Nausea?: Yes | 16 | 17 | 17
  POD1 - Nausea?: No | 28 | 23 | 21
  POD1 - Vomiting?: number analyzed (Participants) | 44 | 40 | 37
  POD1 - Vomiting?: Yes | 1 | 5 | 5
  POD1 - Vomiting?: No | 43 | 35 | 32
  POD1 - Constipation?: number analyzed (Participants) | 44 | 40 | 38
  POD1 - Constipation?: Yes | 19 | 18 | 7
  POD1 - Constipation?: No | 25 | 22 | 31
  POD1 - Difficulty passing urine?: number analyzed (Participants) | 44 | 40 | 37
  POD1 - Difficulty passing urine?: Yes | 11 | 13 | 5
  POD1 - Difficulty passing urine?: No | 33 | 27 | 32
  POD1 - Difficulty concentrating?: number analyzed (Participants) | 44 | 40 | 36
  POD1 - Difficulty concentrating?: Yes | 14 | 18 | 12
  POD1 - Difficulty concentrating?: No | 30 | 22 | 24
  POD1 - Drowsiness/Difficulty Staying Awake?: number analyzed (Participants) | 44 | 40 | 38
  POD1 - Drowsiness/Difficulty Staying Awake?: Yes | 21 | 25 | 21
  POD1 - Drowsiness/Difficulty Staying Awake?: No | 23 | 15 | 17
  POD1 - Lightheaded or dizzy?: number analyzed (Participants) | 44 | 40 | 37
  POD1 - Lightheaded or dizzy?: Yes | 24 | 21 | 18
  POD1 - Lightheaded or dizzy?: No | 20 | 19 | 19
  POD1 - Feeling confused?: number analyzed (Participants) | 44 | 40 | 37
  POD1 - Feeling confused?: Yes | 4 | 8 | 3
  POD1 - Feeling confused?: No | 40 | 32 | 34
  POD1 - Fatigue?: number analyzed (Participants) | 44 | 40 | 38
  POD1 - Fatigue?: Yes | 17 | 23 | 20
  POD1 - Fatigue?: No | 27 | 17 | 18
  POD1 - Itchiness?: number analyzed (Participants) | 44 | 40 | 38
  POD1 - Itchiness?: Yes | 9 | 14 | 13
  POD1 - Itchiness?: No | 35 | 26 | 25
  POD1 - Dry mouth?: number analyzed (Participants) | 44 | 40 | 38
  POD1 - Dry mouth?: Yes | 33 | 36 | 29
  POD1 - Dry mouth?: No | 11 | 4 | 9
  POD1 - Headache?: number analyzed (Participants) | 43 | 40 | 38
  POD1 - Headache?: Yes | 5 | 6 | 3
  POD1 - Headache?: No | 38 | 34 | 35
  POD3 - Nausea?: number analyzed (Participants) | 36 | 36 | 30
  POD3 - Nausea?: Yes | 10 | 12 | 5
  POD3 - Nausea?: No | 26 | 24 | 25
  POD3 - Vomiting?: number analyzed (Participants) | 36 | 36 | 30
  POD3 - Vomiting?: Yes | 2 | 1 | 2
  POD3 - Vomiting?: No | 34 | 35 | 28
  POD3 - Constipation?: number analyzed (Participants) | 36 | 36 | 30
  POD3 - Constipation?: Yes | 21 | 22 | 15
  POD3 - Constipation?: No | 15 | 14 | 15
  POD3 - Difficulty passing urine?: number analyzed (Participants) | 36 | 36 | 30
  POD3 - Difficulty passing urine?: Yes | 5 | 5 | 3
  POD3 - Difficulty passing urine?: No | 31 | 31 | 27
  POD3 - Difficulty concentrating?: number analyzed (Participants) | 36 | 36 | 30
  POD3 - Difficulty concentrating?: Yes | 16 | 19 | 13
  POD3 - Difficulty concentrating?: No | 20 | 17 | 17
  POD3 - Drowsiness/Difficulty Staying Awake?: number analyzed (Participants) | 35 | 36 | 30
  POD3 - Drowsiness/Difficulty Staying Awake?: Yes | 20 | 25 | 18
  POD3 - Drowsiness/Difficulty Staying Awake?: No | 15 | 11 | 12
  POD3 - Lightheaded or dizzy?: number analyzed (Participants) | 36 | 36 | 30
  POD3 - Lightheaded or dizzy?: Yes | 10 | 8 | 8
  POD3 - Lightheaded or dizzy?: No | 26 | 28 | 22
  POD3 - Feeling confused?: number analyzed (Participants) | 36 | 36 | 30
  POD3 - Feeling confused?: Yes | 5 | 4 | 2
  POD3 - Feeling confused?: No | 31 | 32 | 28
  POD3 - Fatigue?: number analyzed (Participants) | 36 | 36 | 30
  POD3 - Fatigue?: Yes | 23 | 24 | 18
  POD3 - Fatigue?: No | 13 | 12 | 12
  POD3 - Itchiness?: number analyzed (Participants) | 36 | 36 | 30
  POD3 - Itchiness?: Yes | 13 | 13 | 10
  POD3 - Itchiness?: No | 23 | 23 | 20
  POD3 - Dry mouth?: number analyzed (Participants) | 36 | 36 | 30
  POD3 - Dry mouth?: Yes | 24 | 19 | 20
  POD3 - Dry mouth?: No | 12 | 17 | 10
  POD3 - Headache?: number analyzed (Participants) | 36 | 36 | 30
  POD3 - Headache?: Yes | 7 | 11 | 10
  POD3 - Headache?: No | 29 | 25 | 20

9. Secondary Outcome: Perioperative Complications - Drain Output
Description: Complications such as: excessive drain output, elevation in creatinine, and the need for transfusions will be identified and recorded
Time Frame: Hospital Stay (1-4 days)
Population: Patient treated Per-Protocol with completed data
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 34 | 38 | 31
mL
  Total Drain output 24H | 270 [135 to 400] | 235 [150 to 348.75] | 240 [160 to 390]
  Total Drain output 48H | 390 [203.75 to 530] | 305 [200 to 515] | 320 [240 to 520]
  Total Drain output 72H | 390 [203.75 to 620] | 335 [200 to 585] | 340 [240 to 520]
  Total Drain output at discharge | 390 [203.75 to 635] | 335 [200 to 605] | 340 [240 to 535]
Statistical Analysis 1: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of Total Drain output at 24H is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.928, Kruskal-Wallis
Statistical Analysis 2: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of Total Drain output at 48H is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.906, Kruskal-Wallis
Statistical Analysis 3: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of Total Drain output at 72H is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.926, Kruskal-Wallis
Statistical Analysis 4: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of Total Drain output at Discharge is the same across the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.934, Kruskal-Wallis

10. Secondary Outcome: Perioperative Complications - Transfusion Rate
Description: as for outcome 9
Time Frame: Hospital Stay (1-4 days)
Population: Patient treated Per-Protocol with completed data
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 44 | 43 | 41
Participants
  No transfusion | 40 | 42 | 41
  Transfusion | 4 | 1 | 0
Statistical Analysis 1: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; Proportion of patient receiving at least 1 transfusion is the same across the 3 arms; Test type: Equivalence — Two-sided; p = 0.078, Chi-squared

11. Secondary Outcome: Days to Walk 50 ft With PT
Description: Days needed to be able to walk 50ft with PT
Time Frame: Hospital Stay (1-4 days)
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 44 | 43 | 41
Participants
  POD0 | 30 | 26 | 24
  POD1 | 11 | 12 | 14
  POD2 and after | 3 | 5 | 3
Statistical Analysis 1: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; Test type: Equivalence — Two-sided 95% confidence interval; p = 0792, Chi-squared

12. Secondary Outcome: Length of Stay
Description: Will record date of discharge
Time Frame: Hospital Stay (1-4 days)
Measure: Mean (Inter-Quartile Range); unit: Hour
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 44 | 43 | 41
Hour | 49.5 [43.25 to 91.25] | 77 [67 to 100] | 70 [47 to 91.5]
Statistical Analysis 1: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of Length of stay in day is the same across these arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.034, Kruskal-Wallis
Statistical Analysis 2: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; The distribution of Length of stay in hour is the same across these arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.030, Kruskal-Wallis

13. Secondary Outcome: Veterans Rand - 12
Description: The Veterans RAND 12 Item Health Survey (VR-12) is a brief, generic, multi-use, self-administered health survey comprised of 12 items. The instrument is primarily used to measure health related quality of life, to estimate disease burden and to evaluate disease-specific benchmarks with other populations. The 12 items in the questionnaire correspond to eight principal physical and mental health domains including general health perceptions; physical functioning; role limitations due to physical and emotional problems; bodily pain; energy-fatigue, social functioning and mental health.. The 12 items are summarized into two scores, a "Physical Health Summary Measure {PCS-physical component score}" and a "Mental Health Summary Measure {MCS-mental component score}". Score range is 0 to 100, higher score denotes a better outcome.
  This score range apply to both PCS and MCS.
Time Frame: pre-operative
Population: Patient treated Per-Protocol with completed follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 43 | 39 | 36
score on a scale
  PCS score | 34.7 (10.8) | 34.2 (10.7) | 34.5 (9.7)
  MCS Score | 43.9 (6.1) | 42.9 (6.7) | 42.0 (7.1)
Statistical Analysis 1: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; Comparison of the PCS score between the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.974, ANOVA
Statistical Analysis 2: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; Comparison of the MCS between the 3 ams; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.444, ANOVA

14. Secondary Outcome: Oswestry Disability Index
Description: The Oswestry Disability Index (ODI) is the most commonly used outcome-measure questionnaire for low back pain in a hospital setting. It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. Thus, for every question not answered, the denominator is reduced by 5. If a patient marks more than one statement in a question, the highest scoring statement is recorded as a true indication of disability.
Time Frame: pre-operative
Population: Patient treated Per-Protocol with pre-operative ODI
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 44 | 41 | 38
percentage | 36.3 (14.3) | 35.4 (11.1) | 40.6 (15.9)
Statistical Analysis 1: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.215, ANOVA

15. Secondary Outcome: Veterans Rand - 12
Description: as for outcome 13
Time Frame: 3 month follow up
Population: Patient treated Per-Protocol with completed follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 31 | 27 | 30
score on a scale
  PCS score | 43.1 (11.8) | 48.7 (8.8) | 42.3 (9.9)
  MCS score | 45.0 (5.3) | 44.3 (6.1) | 45.3 (4.5)
Statistical Analysis 1: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; Comparison PCS score between the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.044, ANOVA
Statistical Analysis 2: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; Comparison MCS score between the 3 arms; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.767, ANOVA

16. Secondary Outcome: Oswestry Disability Index
Description: as for outcome 14
Time Frame: 3 month follow up
Population: patient treated Per-Protocol with completed follow-up
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 38 | 34 | 34
percentage | 22.8 (15.7) | 18.8 (12.9) | 25.0 (13.6)
Statistical Analysis 1: Comparison: IV Ketorolac vs Intravenous (IV) Placebo vs IV Acetaminophen; Test type: Equivalence — Two-sided 95% confidence interval; p = 0.191, ANOVA

17. Secondary Outcome: Return to Work
Description: Record return to work
Time Frame: 3 month follow up
Population: Patient treated Per-Protocol with completed follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 35 | 30 | 33
Participants
  Does not Apply | 9 | 7 | 7
  Early retirement | 1 | 0 | 2
  Complete disability | 3 | 5 | 1
  Lighter job | 3 | 3 | 0
  Original job. part time | 4 | 3 | 3
  Original job, full time | 15 | 12 | 20

18. Secondary Outcome: Veterans Rand - 12
Description: as for outcome 13
Time Frame: 1 year follow up
Population: Patient treated Per-Protocol with completed follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 30 | 28 | 24
score on a scale
  PCS score | 48.1 (11.6) | 47.6 (11.9) | 48.4 (11.1)
  MCS score | 42.8 (5.7) | 45.0 (6.7) | 45.3 (4.4)

19. Secondary Outcome: Oswestry Disability Index
Description: as for outcome 14
Time Frame: 1 year follow up
Population: Patient treated Per-Protocol with completed follow-up
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 36 | 33 | 29
percentage | 16.9 (15.7) | 12.1 (13.3) | 17.8 (14.2)

20. Secondary Outcome: Return to Work
Description: Record return to work
Time Frame: 1 year follow up
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 32 | 29 | 24
Participants
  Does not Apply | 9 | 7 | 3
  Early retirement | 3 | 3 | 4
  Complete disability | 0 | 0 | 1
  Lighter job | 1 | 1 | 0
  Original job, part time | 2 | 2 | 0
  Original job, full time | 17 | 16 | 16

21. Secondary Outcome: Numerical Pain Rating Scale
Description: as for outcome 6
Time Frame: 1 year follow up
Population: Patient treated Per-Protocol with completed follow-up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 27 | 23 | 17
score on a scale
  1-year - Current pain level | 6 [0 to 28] | 7 [0 to 20] | 13 [0.5 to 26.5]
  1-year - Best pain level | 4 [0 to 21] | 0 [0 to 7] | 9 [0 to 22]
  1-year - Worst pain level | 11 [0 to 41] | 8 [0 to 25] | 25 [6.5 to 45.5]

22. Secondary Outcome: Veterans Rand - 12
Description: as for outcome 13
Time Frame: 2 year follow up
Population: Patient treated Per-Protocol with completed follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 26 | 23 | 23
score on a scale
  PCS score | 46.6 (10.7) | 51.2 (9.1) | 51.1 (9.6)
  MCS score | 46.4 (5.8) | 44.5 (4.9) | 46.7 (3.8)

23. Secondary Outcome: Oswestry Disability Index
Description: as for outcome 14
Time Frame: 2 year follow up
Population: Patient treated Per-Protocol with completed follow-up
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 27 | 25 | 25
percentage | 14.7 (14.5) | 11.4 (11.6) | 16.0 (15.1)

24. Secondary Outcome: Return to Work
Description: Record return to work
Time Frame: 2 year follow up
Population: Patient treated Per-Protocol with completed follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 25 | 24 | 26
Participants
  Does not Apply | 5 | 8 | 7
  Early retirement | 5 | 5 | 3
  Complete disability | 0 | 0 | 1
  Lighter job | 0 | 0 | 0
  Original job, part time | 3 | 2 | 0
  Original job, full time | 12 | 9 | 15

25. Secondary Outcome: Numerical Pain Rating Scale
Description: as for outcome 6
Time Frame: 2 year follow up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
Number analyzed (Participants) | 23 | 20 | 22
score on a scale
  2 year - Current pain level | 4 [0 to 41] | 3 [0 to 23.5] | 12.5 [0 to 30.5]
  2 year - Best pain level | 1 [0 to 13] | 0 [0 to 13.25] | 8.5 [1.5 to 19.25]
  2 year - Worst pain level | 13 [0 to 37] | 1.5 [0 to 28.5] | 18 [8 to 50]

ADVERSE EVENTS:
Time Frame: 2-year
Arm/Group | IV Ketorolac | Intravenous (IV) Placebo | IV Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43 | 0/41
Serious Adverse Events (participants affected / at risk) | 10/44 | 9/43 | 11/41
Other Adverse Events (participants affected / at risk) | 40/44 | 40/43 | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Ketorolac (N=44) | Intravenous (IV) Placebo (N=43) | IV Acetaminophen (N=41)
Cardiopulmonary (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 — Hypotension tachycardia hypertension DVT hypoxia palpitations other pulmonary arrhythmia bradycardia pulmonary embolism other cardiopulmonary chest pain cough pleural effusion
cardiovascular (Endocrine disorders) | 0 | 0 | 0 — acute blood loss anemia
Fall (mechanical) (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (syncope) (Injury, poisoning and procedural complications) | 0 | 0 | 0
Gastrointestinal (Gastrointestinal disorders) | 0 | 0 | 0 — nausea nausea/vomiting distention constipation ileus diarrhea other gastrointestinal pain abdominal pain
Implant-related (Surgical and medical procedures) | 1 | 2 | 0
Infection (Infections and infestations) | 0 | 2 | 0 — UTI Superficial infection deep infection
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 6 | 2 | 1 — leg pain gout back pain knee pain hip pain hand pain neck pain arthritis foot pain fracture carpal tunnel shoulder pain low back pain
Neurologic (Nervous system disorders) | 3 | 5 | 10 — Radiculopathy Sensory deficit motor deficit/weakness cervical radiculopathy spasm mental status change Radiculopathy cervical Sensory deficit
Operative (Surgical and medical procedures) | 0 | 0 | 0 — Dural Tear Monitoring anomaly (SSEP) Monitoring Anomaly vascular injury
Radiographic (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 — adjacent segment degeneration pseudarthrosis
Renal (Renal and urinary disorders) | 0 | 0 | 1 — oliguria urinary retention hematuria Electrolyte imbalance
Vascular (Vascular disorders) | 0 | 0 | 0 — edema
Wound (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 — prolonged drainage seroma swelling redness pain
Other (General disorders) | 1 | 0 | 1 — ABLA, Fever, lightheaded/dizzy, pruritis, headache, adhesive reaction, rash, cancer, trigger finger, sore throat, dermatological, tear in the throat, elevated liver enzymes, sinusitis, transaminitis, rhinitis, hearing, bone quality, hyperglycemia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Ketorolac (N=44) | Intravenous (IV) Placebo (N=43) | IV Acetaminophen (N=41)
cardiopulmonary (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 8 — Hypotension tachycardia hypertension DVT hypoxia palpitations other pulmonary arrhythmia bradycardia pulmonary embolism other cardiopulmonary chest pain cough pleural effusion
cardiovascular (Endocrine disorders) | 0 | 0 | 1 — acute blood loss anemia
fall (mechanical) (Injury, poisoning and procedural complications) | 1 | 2 | 2
fall (syncope) (Injury, poisoning and procedural complications) | 1 | 0 | 1
gastrointestinal (Gastrointestinal disorders) | 15 | 15 | 8 — nausea nausea/vomiting distention constipation ileus diarrhea other gastrointestinal pain abdominal pain
implant-related (Surgical and medical procedures) | 0 | 0 | 0
infection (Infections and infestations) | 4 | 0 | 0 — UTI Superficial infection deep infection
musculoskeletal (Musculoskeletal and connective tissue disorders) | 13 | 12 | 6 — leg pain gout back pain knee pain hip pain hand pain neck pain arthritis foot pain fracture carpal tunnel shoulder pain low back pain
neurologic (Nervous system disorders) | 26 | 18 | 32 — Radiculopathy Sensory deficit motor deficit/weakness cervical radiculopathy spasm mental status change Radiculopathy cervical Sensory deficit
operative (Surgical and medical procedures) | 1 | 4 | 0 — Dural Tear Monitoring anomaly (SSEP) Monitoring Anomaly vascular injury
radiographic (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 — adjacent segment degeneration pseudarthrosis
renal (Renal and urinary disorders) | 4 | 13 | 8 — oliguria urinary retention hematuria Electrolyte imbalance Other
vascular (Vascular disorders) | 0 | 3 | 4 — edema
wound (Skin and subcutaneous tissue disorders) | 9 | 1 | 2 — prolonged drainage seroma swelling redness pain
other (General disorders) | 23 | 23 | 14 — ABLA, Fever, lightheaded/dizzy, pruritis, headache, adhesive reaction, rash, cancer, trigger finger, sore throat, dermatological, tear in the throat, elevated liver enzymes, sinusitis, transaminitis, rhinitis, hearing, bone quality, hyperglycemia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT02700451/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT02700451/ICF_001.pdf